CLINICAL TRIAL: NCT05598307
Title: The Anesthetic and Analgesic Effects of Intravenous Magnesium Sulphate in Elective Laparoscopic Cholecystectomy
Brief Title: A Study of the Effects of Intravenous Magnesium Sulphate on Anaesthesia and Analgesia in Elective General Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13/22-09-2021
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Nociceptive; Analgesia; Magnesium
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Nociceptive Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- magnesium bolus (Active Comparator): A bolus dose of magnesium of 40 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Followingly, normal saline will be administered at a rate of 20 mL/h
  Interventions: Drug: magnesium bolus followed by normal saline infusion
- magnesium bolus and magnesium infusion (Active Comparator): A bolus dose of magnesium of 40 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Followingly, 10 mg/kg/h of magnesium will be administered intraoperatively diluted in a 60 mL syringe and administered at a rate of 20 mL/h
  Interventions: Drug: magnesium bolus followed by magnesium infusion
- placebo (Placebo Comparator): 100 mL of normal saline will be administered within 10 minutes preoperatively. Followingly, normal saline will be administered at a rate of 20 mL/h
  Interventions: Drug: normal saline bolus followed by normal saline infusion

INTERVENTIONS:
Drug: magnesium bolus followed by normal saline infusion — a bolus dose of magnesium will be followed by normal saline infusion
  Arms: magnesium bolus
Drug: magnesium bolus followed by magnesium infusion — a bolus dose of magnesium will be followed by a magnesium infusion
  Arms: magnesium bolus and magnesium infusion
Drug: normal saline bolus followed by normal saline infusion — a bolus of normal saline will be followed by normal saline infusion
  Arms: placebo

SUMMARY:
The aim of this double-blind randomized study will be to evaluate the effect an intravenous infusion of magnesium has on recovery outcomes after elective laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Magnesium consists one of the most important electrolytes of the human body, producing effects in various systems, one of them being the central nervous system. It has been shown that the administration of intravenous magnesium sulphate during anesthesia can significantly reduce the requirements for anaesthetic and analgesic agents, perioperatively, and improve the quality of post anesthetic recovery. The present study will examine the effect of administering intravenous magnesium sulphate during anesthesia in patients undergoing elective laparoscopic cholecystectomy surgery. This is a single centre, double-blinded, randomised controlled trial in an adult population, taking place in a tertiary medical centre in Athens. The study consists of three comparison groups of equivalent population, produced by double blinded randomisation. Each comparison arm will be administered a different regimen of magnesium sulphate/placebo. During the perioperative time, depth of anaesthesia will be monitored using the Bispectral Index, (BIS™) and the nociceptive level with nociception level index (NOL®). Dosing of the anaesthetic agent, desflurane, as well as of the analgesic medication, remifentanil, will be adjusted according to the prior indices. Patients included in the study will be monitored in the PACU and the surgical ward for the first 24 hours, postoperatively. Primary outcomes include the requirements for anaesthetic and analgesic agents, time to emergence, time to extubation, time to recovery, quality of recovery variables, pain scores during the first 24 hours and adverse effects and/or complications of magnesium administration. Ethical approval for this trial has been granted by the Ethics Committee of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patents
* American Society of Anesthesiologists (ASA) class I-III
* elective laparoscopic cholecystectomy

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* systematic use of analgesic agents preoperatively
* chronic pain syndromes preoperatively
* neurological or psychiatric disease on treatment
* pregnancy
* severe hepatic or renal disease
* drug or alcohol abuse
* language or communication barriers lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU) | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

OTHER OUTCOMES:
time to first request for analgesia | during stay in Post-Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  the time for the first patient request for analgesia will be noted
morphine consumption in Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  mg of morphine requested during patient PACU stay
pethidine consumption in the first 48 hours | 48 hours postoperatively
  patients will be followed for cumulative pethidine consumption for 48 hours postoperatively
remifentanil requirement during surgery | intraoperatively
  dose of required remifentanil intraoperatively to maintain systolic arterial blood pressure and heart rate within the 20% of baseline value
number of participants experiencing side effects intraoperatively | intraoperatively
  patients will be monitored for side-effects of the administered agents intraoperatively
number of participants experiencing side effects postoperatively | 48 hours postoperatively
  patients will be monitored for side-effects of the administered agents postoperatively
time to emergence | end of operation, approximately 1 hour after start of surgery
  time from desflurane discontinuation to first patient response (eye opening)
time to extubation | end of operation, approximately 1 hour after start of surgery
  time from desflurane discontinuation to tracheal extubation
duration of nociception level<25 intraoperatively | intraoperatively
  nociception level (NOL) is a device that measures the status of analgesia intraoperatively. Levels<25 suggest adequate intraoperatively analgesia

CONTACTS AND LOCATIONS:
Overall Officials: KASSIANI THEODORAKI, PhD, DESA, Principal Investigator — Aretaieion University Hospital, National and Kapodistrian University of Athens, Greece
Locations (1):
- General Hospital of Nikea, Piraeus, Attiki, Greece, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haryalchi K, Abedinzade M, Khanaki K, Mansour Ghanaie M, Mohammad Zadeh F. Whether preventive low dose magnesium sulphate infusion has an influence on postoperative pain perception and the level of serum beta-endorphin throughout the total abdominal hysterectomy. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):384-390. doi: 10.1016/j.redar.2016.11.009. Epub 2017 Feb 14. English, Spanish. PMID 28214095